CLINICAL TRIAL: NCT01455168
Title: Prospective Study to Examine the Efficacy of a Capsular Tension Ring (CTR) in Preventing Anterior Capsule Shrinkage After Cataract Surgery in Exfoliation Syndrome (XFS) With no Zonular Weakness
Brief Title: Efficacy of a Capsular Tension Ring in Preventing Anterior Capsule Shrinkage After Cataract Surgery in Exfoliation Syndrome
Acronym: Effect of CTR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Occupational and Environmental Health (Other)
Responsible Party: Principal Investigator, Yukinori Harada, Assistant Professor, University of Occupational and Environmental Health
Other Study IDs: H23-75; H23-75 (Other: Institutional Review Board of UOEH)
Record Dates: First submitted 2011-09-24; First posted 2011-10-19 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Cataract With Exfoliation Syndrome
Keywords: anterior capsule shrinkage; capsular tension ring; exfoliation syndrome; phacoemulsification and aspiration
MeSH Terms: conditions — Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- No treatment: Capsular tension ring is not used in the group.
- CTR simply implanted: Capsular tension ring is simply implanted in the group.
- CTR with the eyelets closed: Capsular tension ring is implanted and closed by tying both eyelets in the group.

SUMMARY:
The purpose of this study is to examine the efficacy of a capsular tension ring (CTR) in preventing anterior capsule shrinkage after cataract surgery in exfoliation syndrome (XFS) with no zonular weakness. The eyes with XFS undergo phacoemulsification and aspiration (PEA) with an intraocular lens (IOL) implantation. All operations are performed by a single surgeon. No eyes with either ectopia lentis or phacodonesis are included. There are three groups; CTR is not used in group A, CTR is simply implanted in group B, and CTR is implanted and closed by tying both eyelets in group C. The areas of continuous curvilinear capsulorhexis (CCC) are calculated, and both the time-course change and the comparison among the 3 groups are tested.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with exfoliation syndrome are included.

Exclusion Criteria:

* Eyes with either ectopia lentis or phacodonesis are excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients with cataract and exfoliation syndrome
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2004-09; Primary Completion 2006-05 (Actual); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of a Capsular Tension Ring in Preventing Anterior Capsule Shrinkage after Cataract Surgery in Exfoliation Syndrome | 3 years
  The vertical diameters (A mm) and horizontal diameters (B mm) of the postoperative capsulorhexis opening were measured using the scale of a Haag-Strait slit lamp. The area of the rhexis is equal to πAB/4 mm2. The measurements are taken on day one (baseline), and thereafter at each weeks postoperatively. The statistical analyses are used for time-course changes in each group, and for the area among the three groups on the same postoperative period. For this study, the percent change is calculated based on the ratio of the area at each measurement in comparison to the initial value.
Efficacy of a Capsular Tension Ring in Preventing Anterior Capsule Shrinkage after Cataract Surgery in Exfoliation Syndrome | 3 years
  The vertical diameters (A mm) and horizontal diameters (B mm) of the postoperative capsulorhexis opening are measured using the scale of a Haag-Strait slit lamp. The area of the rhexis is equal to πAB/4 mm2. The measurements are taken on day one (baseline), and thereafter at each weeks postoperatively. The statistical analyses are used for time-course changes in each group, and for the area among the three groups on the same postoperative period. For this study, the percent change is calculated based on the ratio of the area at each measurement in comparison to the initial value.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Occupational and Environmental Health, Kitakyushu, Fukuoka, Japan